CLINICAL TRIAL: NCT01509612
Title: Prospective, Randomized, Placebo-controlled, Double-blind, Multicenter Study Evaluating Quality of Life in Patients With Advanced Malignant Lung Tumors With or Without "add-on" Homeopathy
Brief Title: Additive Homeopathy in Cancer Patients
Acronym: HIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Frass, Principal Investigator, Prof. Dr., Director, Outpatient Unit Homeopathy in tumor patients, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 5
Record Dates: First submitted 2012-01-07; First posted 2012-01-13 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Malignant Tumors
Keywords: cancer; additive homeopathy; patients with advanced malignant tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Additive homeopathy in cancer patients (Active Comparator): Lung cancer patients receiving conventional chemo- and/or radiation therapy receive additive classical homeopathy with homeopathic globules
  Interventions: Drug: Additive classical homeopathy
- Additive homeopathic placebo globules (Placebo Comparator): Lung cancer patients receiving conventional chemo- and/or radiation therapy receive homeopathic placebo globules
  Interventions: Drug: Homeopathic Placebo globules
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Additive classical homeopathy — Homeopathic remedies every 2 to 3 months
  Other Names: Classical homeopathic remedies
  Arms: Additive homeopathy in cancer patients
Drug: Homeopathic Placebo globules — Homeopathic placebo globules every 2 to 3 months
  Other Names: Homeopathic Placebo globules looking identical to verum
  Arms: Additive homeopathic placebo globules

SUMMARY:
The investigators aim to investigate the validity of their previous results in a randomized prospective, placebo-controlled, double-blind, multicenter controlled evaluation of questionnaires in patients with advanced malignant tumors. The investigators plan to compare the treatment outcome (quality of life and survival) in tumor patients, receiving standard or "add-on" homeopathic treatment.

The null hypothesis is that "add-on" homeopathic treatment does not create a benefit for cancer patients. In addition the investigators evaluate survival time.

DETAILED DESCRIPTION:
The EORTC-QLQ-C30, SF-36 as well as a VAS scale for subjective well-being will be filled out by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Clinical diagnosis of advanced tumor stages of non small-cell lung carcinoma (NSCLC) IIIB, IIIC, IV.

Exclusion Criteria:

* sensitizing mutation of the EGFR gene or translocation of the ALK gene
* refusal to sign informed consent
* pregnancy
* hematological, hepatic, or renal pathology
* coronary heart disease
* history of secondary tumor
* major surgery within 4 weeks prior to study entry
* active infection and symptomatic peripheral neuropathy
* central nervous system metastases unless the metastases were treated and stable
* active autoimmune disease
* use of systemic immunosuppressive treatment
* use of systemic treatment during the previous 2 years
* active interstitial lung disease, or a history of pneumonitis for which glucocorticoids were prescribed
* previous systemic therapy for metastatic disease or previous irradiation
* use of any complementary and/or alternative therapy, including homeopathy other than the research treatment during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, Prof. Dr., Principal Investigator — Medical University Vienna
Locations (1):
- Michael Frass, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frass M, Lechleitner P, Grundling C, Pirker C, Grasmuk-Siegl E, Domayer J, Hochmair M, Gaertner K, Duscheck C, Muchitsch I, Marosi C, Schumacher M, Zochbauer-Muller S, Manchanda RK, Schrott A, Burghuber O. Homeopathic Treatment as an Add-On Therapy May Improve Quality of Life and Prolong Survival in Patients with Non-Small Cell Lung Cancer: A Prospective, Randomized, Placebo-Controlled, Double-Blind, Three-Arm, Multicenter Study. Oncologist. 2020 Dec;25(12):e1930-e1955. doi: 10.1002/onco.13548. Epub 2020 Nov 7. PMID 33010094
- See also: Related info — http://www.homeopathicresearch.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from February 2012 to July 2017
Pre-assignment Details: Screened participants were excluded from participation in the study when mutations had been observed, these were treated as screening failures and not included in the trial (= not randomized, n=8).
Groups:
- Homeopathic Placebo Globules: Cancer patients received homeopathic placebo remedies
- Additive Classical Homeopathy in Cancer Patients: Lung cancer patients receive additive classical homeopathy with homeopathic remedies
- No Intervention Group: The patients in this group received no intervention
Period: Overall Study
Arm/Group | Homeopathic Placebo Globules | Additive Classical Homeopathy in Cancer Patients | No Intervention Group
Started | 47 | 51 | 52
Completed | 47 | 51 | 52
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Intervention: Lung cancer patients receiving conventional chemo- and/or radiation therapy but neither homeopathic remedies nor homeopathic placebo globules, these patients served as a non-intervention control group
- Total: Total of all reporting groups
Arm/Group | Additive Homeopathy in Cancer Patients | Additive Homeopathic Placebo Globules | No Intervention | Total
Number analyzed (Participants) | 51 | 47 | 52 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.8) | 62.5 (8.9) | 63.9 (9.1) | 63.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 24 | 69
  Male | 26 | 27 | 28 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 51 | 47 | 52 | 150
EORTC-QLQ-C30 [Mean (Standard Deviation); unit: units on a scale from 1 to 4] — At baseline the quality of life questionnaire (EORTC-QLQ-C30) was completed by all participating subjects receiving placebo or homeopathy Population: The quality of life assessment was done in the two intervention groups (homeopathy or placebo), but was not done in control patients who received no intervention.
  Therefore, no data are presented for the "No Intervention" group.
  units on a scale from 1 to 4
    number analyzed (Participants) | 51 | 47 | 0 | 98
    (all) | 46.6 (25.8) | 51.2 (28.0) |  | 48.8 (26.8)

OUTCOME MEASURES:

1. Primary Outcome: EORTC-QLQ-C30 Score
Description: Quality of life was evaluated by using the Global Health Status assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC-QLQ-C30), which was completed by participants throughout the study.
  The score of the scale ranges from 0-100, where high values mean good health status, while lower values indicate poor health status.
Time Frame: baseline and at 18 weeks
Population: Data not collected for the no Intervention Group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- No Intervention Group: Lung cancer patients received conventional anti-cancer therapy, but neither homeopathic remedies nor homeopathic placebo globules. Data not collected for the no Intervention Group.
Arm/Group | Homeopathic Placebo Globules | Additive Classical Homeopathy in Cancer Patients | No Intervention Group
Number analyzed (Participants) | 47 | 51 | 0
score on a scale | 51.2 (28.0) | 46.6 (25.8) |
Statistical Analysis 1: Comparison: Homeopathic Placebo Globules vs Additive Classical Homeopathy in Cancer Patients; Test type: Superiority; p = 0.397, t-test, 2 sided

2. Secondary Outcome: Survival
Description: Survival was assessed by chart review, at every study visit (every 9 weeks throughout the trial), and by information of the central mortality registry of Austria
Time Frame: 2 years for the individual patient (=whole study duration)
Measure: Number; unit: participants
Groups:
- No Intervention: No homeopathic or placebo intervention
Arm/Group | Additive Homeopathy in Cancer Patients | Additive Homeopathic Placebo Globules | No Intervention
Number analyzed (Participants) | 51 | 47 | 52
participants | 23 | 11 | 7
Statistical Analysis 1: Comparison: Additive Homeopathy in Cancer Patients vs Additive Homeopathic Placebo Globules; Only those groups were compared who received an intervention; Test type: Superiority; p = 0.02, Chi-squared

ADVERSE EVENTS:
Time Frame: The study for each participant lasted 24 months
Description: The adverse events reporting in this study differed from the definition of clinicaltrials.gov.
  Treatment-related (serious) and non-treatment-related adverse events have been reported.
  No severe treatment-related (serious) or non-treatment-related adverse event has been identified attributed to the study medication.
Groups:
- Homeopathic Placebo Globules: Cancer patients received homeopathic placebo remedies.
  Treatment emergent and serious adverse events were documented.
- Additive Classical Homeopathy in Cancer Patients: Lung cancer patients receive additive classical homeopathy with homeopathic remedies
  Treatment emergent and serious adverse events were documented.
- No Intervention Group: Patients received no intervention.
  Treatment emergent and serious adverse events were documented.
Arm/Group | Homeopathic Placebo Globules | Additive Classical Homeopathy in Cancer Patients | No Intervention Group
All-Cause Mortality (participants affected / at risk) | 11/47 | 23/51 | 7/52
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 0/47 | 0/51 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT01509612/Prot_SAP_001.pdf